CLINICAL TRIAL: NCT02393040
Title: A Prospective Double Blind, Placebo Controlled Study to Assess the Efficacy of Platelet-Rich Plasma on the Treatment of Androgenetic Alopecia
Brief Title: Study to Assess Efficacy of Platelet-Rich Plasma in Androgenetic Alopecia
Acronym: PRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Rubina Alves, Specialist in Dermatology, M.D., Universitat Internacional de Catalunya
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: UICatalunya
Record Dates: First submitted 2015-03-03; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Androgenetic Alopecia; Alopecia; Hair Loss
Keywords: Alopecia; Androgenetic Alopecia; Alopecia, Male Pattern; Hair loss; Platelet-Rich Plasma; Alopecia, Female Pattern; placebo; double-blind
MeSH Terms: conditions — Alopecia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRP/Saline (Experimental): PRP/Saline
  Briefly, for PRP preparation, approximately 18 mL of blood from each patient is drawn into a tube containing 3,8 % sodium citrate. The tubes were centrifuged at 450 g for 8 minutes, resulting in three basic layers: an erythrocyte layer at the bottom of the tube, a PRP layer in the middle, and a platelet-poor plasma (PPP) layer at the top of the tube. After removing the platelet-poor plasma (PPP) layer, the PRP is obtained, activated with 10 % calcium chloride.
  In the same patient, PRP will be injected to half-head and in the other half-head will be injected with saline solution (placebo).
  This study includes 4 visits: 3 visits (with 1-month interval) and 1 visit of follow-up (month 6).
  Interventions: Other: PRP/Saline

INTERVENTIONS:
Other: PRP/Saline — PRP/Saline: Two groups were defined: group A and group B. Group A received treatment with PRP on the right half-head and placebo on the left half-head while group B received administration of PRP on left half-head and placebo on the right half-head.
  Same patient will be injected with PRP and a saline solution. Each patient will be injected on half-head.
  Other Names: PRP; androgenetic alopecia; alopecia; hair Loss; placebo; saline

SUMMARY:
The purpose of this study is to determine the efficacy of treatment with Platelet-rich plasma on Androgenetic alopecia (compared with placebo), between six months and baseline.

DETAILED DESCRIPTION:
Androgenetic alopecia (AGA) is a non-scarring patterned alopecia, multifactorial and a genetic determined skin condition. This pathology is one of the most common forms of progressive hair loss. It's an increasingly frequent complaint of dermatology clinic patients and has a high impact psychologically.

The onset of AGA is gradual and when this pathology progresses, the anagen phase shortens and the telogen phase remains constant. As a result, more hairs are in the telogen phase, and the patient may notice an increase in hair shedding. This area varies from patient to patient and is usually most marked at the vertex in men while women with androgenetic alopecia generally lose hair diffusely over the crown. The incidence and prevalence of AGA increases with age.

Topical minoxidil and oral finasteride are the gold standard therapies for AGA and the only two drugs currently that have US Food and Drug Administration (FDA)-approved indications for the treatment of androgenetic alopecia. Minoxidil and finasteride are known to be effective medical treatments in AGA, especially during the initial grades.

PRP is a plasma concentrate reaped from the patient's whole blood that comprises predominantly platelets. Numerous growth factors (GFs) are present within platelet α granules. Some of the most important of these include platelet-derived growth factor (PDGF), transforming growth factor-beta (TGF-β), vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), and insulin-like growth factor (IGF). This GFs stimulate cell proliferation and differentiation.

PRP was identified as having a beneficial effect on bone grafting with applications in oral and maxillofacial surgery, orthopedic and cardiac surgery. More recently, increasing interest is seen in the application of PRP in dermatology, for example, tissue regeneration, wound healing such and fat grafting. It has also been shown to promote hair survival and growth, both in vitro and in vivo.

The production of autologous PRP involves extraction of a specific volume of the patient's whole blood, which is then placed in an automated centrifuge to separate the layers of whole blood by their specific weight into 3 separate layers: (1) platelet-poor plasma, (2) platelet-rich plasma and (3) red blood cells.

The patients were divided into two groups (A and B): group A received treatment with PRP on the right half-head and the placebo on the left half-head, whereas group B received treatment with PRP on the left half-head and the placebo on the right half-head.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years and < 65 years
* Male patients with a clinical diagnosis of AGA (stage II to V according to the Hamilton-Norwood Scale)
* Female patients with a clinical diagnosis of AGA (stage I to III according to Ludwig Classification)

Exclusion Criteria:

* Patients with other types of alopecia, other than AGA
* Fasting < 3h prior of each injection
* Use of nonsteroidal anti-inflammatory drugs one week before treatment.
* Platelet count < 150 000 μL
* Alterations of coagulation
* Heavy smokers (> 20 cigarettes/day)
* Medications: anticoagulants/ acetylsalicylic acid
* Patient unable to accomplishing all fases of treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Determine the treatment efficacy by measuring hair regrowth score for each side of scalp. | 6 months

SECONDARY OUTCOMES:
Determine the treatment efficacy by measuring hair density for each side of scalp | 6 months
  Determine the treatment efficacy by measuring mean hair density for each side of scalp using the trichogram analysis.
Determine the treatment efficacy by measuring anagen/telogen ratio for each side of scalp | 6 months
  Determine the treatment efficacy by measuring anagen/telogen ratio for each side of scalp using the trichogram analysis.
Global photographs of three areas of the scalp (evaluation of hair growth will be assessed by comparison of standardized images) | 6 months
  The evaluation of hair growth will be assessed by comparison of standardized images between baseline and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Alves, M.D., Principal Investigator — Specialist Dermatology, Universitat Internacional Catalunya; Ramon Grimalt, M.D.; PhD, Study Director — Prof. Dermatology, Universitat Internacional Catalunya
Locations (1):
- Universitat Internacional Catalunya, Barcelona, Barcelona, Spain